CLINICAL TRIAL: NCT01200277
Title: A Randomised Sham Controlled Trial of Vertebroplasty for Painful Acute Osteoporotic Vertebral Fractures
Brief Title: A Trial of Vertebroplasty for Painful Acute Osteoporotic Vertebral Fractures
Acronym: VertosIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Responsible Party: Principal Investigator, Willem Jan van Rooij, WJ van Rooij, St. Elisabeth Ziekenhuis., Elisabeth-TweeSteden Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EZTilburg1
Record Dates: First submitted 2010-09-07; First posted 2010-09-13 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Osteoporosis; Vertebral Fracture
Keywords: osteoporosis; vertebral fracture; vertebroplasty; percutaneous
MeSH Terms: conditions — Osteoporosis; Spinal Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- vertebroplasty (Experimental): Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine). For the vertebroplasty procedure, 11-gauge or 13-gauge needles are passed into the central aspect of the target vertebra or vertebrae. Bone cement is prepared on the bench and injected under constant fluoroscopy into the vertebral body. Injection is stopped when the cement reaches to the posterior aspect of the vertebral body or leaks into an extraosseous space, such as the intervertebral disk or an epidural or paravertebral vein.
  Interventions: Procedure: percutaneous vertebroplasty
- sham procedure (Sham Comparator): Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine). During the sham intervention, verbal and physical cues, such as pressure on the patient's back, are given, and the bone cement is prepared to simulate the odor associated with mixing of polymethacrylate , but the needle is not placed and cement is not injected.
  Interventions: Procedure: sham procedure

INTERVENTIONS:
Procedure: percutaneous vertebroplasty — Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine. For the vertebroplasty procedure, 11-gauge or 13-gauge needles are passed into the central aspect of the target vertebra or vertebrae. Bone cement is prepared on the bench and injected under constant fluoroscopy into the vertebral body. Injection is stopped when the PMMA reaches to the posterior aspect of the vertebral body or leaks into an extraosseous space, such as the intervertebral disk or an epidural or paravertebral vein.
  Arms: vertebroplasty
Procedure: sham procedure — Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine. During the sham intervention, verbal and physical cues, such as pressure on the patient's back, are given, and the methacrylate monomer is opened to simulate the odor associated with mixing of cement, but the needle is not placed and cement is not injected.
  Arms: sham procedure

SUMMARY:
The standard care in patients with a painful osteoporotic vertebral compression fracture (VCF) is conservative therapy. Percutaneous vertebroplasty (PV), is a new minimally invasive technique for pain treatment in which bone cement is injected in the fractured vertebra. Recent RCTs provide conflicting results: two sham-controlled studies show no benefit of PV while an unmasked but controlled RCT found significantly better pain relief after PV at acceptable costs.

DETAILED DESCRIPTION:
Objectives To evaluate the efficacy of bone cement injection in PV for patients with acute painful osteoporotic compression fractures, as compared with a simulated placebo procedure without injection of bone cement. We hypothesize that patients who had undergone PV would report less pain at 1 day, 1 week and 1, 3, 6 and 12 months (the primary outcomes) than those in the sham control group.

Study design VERTOS IV is a multicenter RCT concerning the treatment of patients with a painful osteoporotic VCF. Patients are recruited on the Radiology departments of the participating hospitals and randomized to PV or a simulated procedure. Upon obtaining informed consent an independent central telephone operator completes the randomisation procedure, using a computer program. The maximum allowed unbalance (block size) is six, with a maximum sample size of 84 for each participating centre. A total of 180 patients will be enrolled, 90 in each group. This is based on the assumption of a 1.5 point difference in pain relief (VAS Score) and a 20% withdrawal rate (α=0.05 and β=0.20, 7 measurement points). The enrolment of patients will take place in four centres in The Netherlands: St. Elisabeth Ziekenhuis in Tilburg, Catharina Ziekenhuis in Eindhoven, Medisch Spectrum Twente in Enschede and Albert Schweitzer Ziekenhuis in Dordrecht. Randomization will start January 2011 with an expected completion of enrolment by January 2013. There is a one-year follow-up, with the possibility of an extended follow-up at two years.

The overall Institutional Review Board is approval is obtained at the St. Elisabeth Hospital in Tilburg. In addition, each participating centre will obtain a local Institutional Review Board Approval. This study is registered at ClinicalTrials.gov., NCT01200277.

Osteoporosis- and pain medication All patients receive osteoporosis medication, such as bisphosphonates together with supplemental calcium and vitamin D. Pain medication demanded by the patient is recorded. Analgesics are classified following the WHO classification: (1) Paracetamol (acetaminophen), (2) Tramadol, (3) Tramadol and Paracetamol, (4) Morphine. Non Steroid Anti Inflammatory Drugs (NSAID) are only prescribed if patients are intolerant for opiate-derivatives or when already used. Corrections in dose and classification of pain medication are made if necessary.

Clinical follow-up An experienced nurse-practitioner requests patients to fill out a standard questionnaire before and at 1 day, 1 week, and 1, 3, 6 and 12 months after the procedure. The questionnaire consist of the VAS score and questions about use of pain medication, pain location, and pain type. The VAS score is a pain score ranging from 0 (no pain) to 10 (worst pain ever. Other medical treatment and visits to alternative medical specialists, GP's and physical therapists are recorded and compared between groups. Secondary outcomes are back pain related disability and QOL as measured with the Roland Morris Disability (RMD) Questionnaire and the Questionnaire of the European Foundation for Osteoporosis (Qualeffo), respectively. The Qualeffo is developed specifically for patients with osteoporosis. This questionnaire consists of 41 questions about: pain, physical function, social function, general health perception, and mental function. The Qualeffo score ranges from 0 (best quality of life) to 100 (worst quality of life). This questionnaire will be completed at five measurement moments (before and at 1, 3, 6, and 12 months after the procedure). The RMD questionnaire is a disability questionnaire that measures the functional status of patients with back pain. The RMD will be completed at all measurement points. All patients visit the internist at 1,3,6 and 12 months follow-up. All patients receive a pain diary. Patients are asked to fill out the VAS score and use of analgesics is recorded on a daily basis during the first month after randomization.

Sample size considerations Assuming a 1.5 point difference in pain relief as measured by VAS score and a withdrawal rate of 20% (α=0.05 and β=0.20, 7 measurement points), a total of 180 patients will be enrolled, 90 in each group.

Statistical analysis The data will be analysed according to the intention-to-treat principle. Standard statistical techniques will be used to describe characteristics of patients in both groups. We will compare baseline characteristics in the two treatment groups and if incomparability appears, we will in secondary analysis adjust for differences. The primary outcome, significant pain relief will be compared with the analysis of variance for repeated measures. If adjustment for possible baseline incomparability is needed, analysis of covariance will be done. Since we expect the difference between the two groups will particularly become evident at 3, 6 and 12 months, the analysis will also be performed at these time points.

ELIGIBILITY:
Inclusion Criteria:

* VCF on X-ray of the spine (minimal 15% loss of height)
* level of VCF Th5 or lower
* back pain ≤ 6 weeks at time of X-ray
* ≥ 50 years of age
* bone edema on MRI of the fractured vertebral body
* focal tenderness on VCF level
* decreased bone density T-scores ≤ -1

Exclusion Criteria:

* severe cardio-pulmonary condition
* untreatable coagulopathy
* systemic or local infection of the spine (osteomyelitis, spondylodiscitis)
* suspected alternative underlying disease (malignancy)
* radicular and/or cauda compression syndrome
* contra-indication for MRI

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
pain relief | 12 months
  Primary outcome will be pain relief at 1 day, 1 week, and 1,3, 6 and 12 months. The questionnaire consist of the VAS score and questions about use of pain medication, pain location, and pain type. Other medical treatment and visits to alternative medical specialists, GP's and physical therapists are recorded and compared between groups. Patients are asked to fill out the VAS score and use of analgesics is recorded on a daily basis during the first month after randomization.

SECONDARY OUTCOMES:
back pain related disability | 0, 1day, 1 week, 1,3,6,12 months
  Back pain related disability as measured with the Roland Morris Disability (RMD) Questionnaire. The Qualeffo is developed specifically for patients with osteoporosis. This questionnaire consists of 41 questions about: pain, physical function, social function, general health perception, and mental function. The RMD questionnaire is a disability questionnaire that measures the functional status of patients with back pain.
Quality of Life | 1 week, 1,3,6,12 months
  QOL as measured with the Questionnaire of the European Foundation for Osteoporosis (Qualeffo). The Qualeffo is developed specifically for patients with osteoporosis. This questionnaire consists of 41 questions about: pain, physical function, social function, general health perception, and mental function. The Qualeffo score ranges from 0 (best quality of life) to 100 (worst quality of life). This questionnaire will be completed at five measurement moments (before and at 1, 3, 6, and 12 months after the procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Willem Jan van Rooij, PhD, Study Director — St. Elisabeth Ziekenhuis; Paul N Lohle, PhD, Principal Investigator — St Elisabeth Ziekenhuis; Jolanda De Vries, PhD, Study Director — St Elisabeth Ziekenhuis
Locations (4):
- Netherlands (4):
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - St. Elisabeth Ziekenhuis, Tilburg

REFERENCES:
- [Derived] Firanescu CE, de Vries J, Lodder P, Schoemaker MC, Smeets AJ, Donga E, Juttmann JR, Klazen CAH, Elgersma OEH, Jansen FH, van der Horst I, Blonk M, Venmans A, Lohle PNM. Percutaneous Vertebroplasty is no Risk Factor for New Vertebral Fractures and Protects Against Further Height Loss (VERTOS IV). Cardiovasc Intervent Radiol. 2019 Jul;42(7):991-1000. doi: 10.1007/s00270-019-02205-w. Epub 2019 Apr 2. PMID 30941490
- [Derived] Firanescu CE, de Vries J, Lodder P, Venmans A, Schoemaker MC, Smeets AJ, Donga E, Juttmann JR, Klazen CAH, Elgersma OEH, Jansen FH, Tielbeek AV, Boukrab I, Schonenberg K, van Rooij WJJ, Hirsch JA, Lohle PNM. Vertebroplasty versus sham procedure for painful acute osteoporotic vertebral compression fractures (VERTOS IV): randomised sham controlled clinical trial. BMJ. 2018 May 9;361:k1551. doi: 10.1136/bmj.k1551. PMID 29743284
- [Derived] Firanescu C, Lohle PN, de Vries J, Klazen CA, Juttmann JR, Clark W, van Rooij WJ; VERTOS IV study group. A randomised sham controlled trial of vertebroplasty for painful acute osteoporotic vertebral fractures (VERTOS IV). Trials. 2011 Apr 5;12:93. doi: 10.1186/1745-6215-12-93. PMID 21466679